CLINICAL TRIAL: NCT05235724
Title: Open-label 12-week Longitudinal Exploratory Study to Assess Reliability/Feasibility of Using Emerald Touchless Sensor for Scratching and Sleep Quantification in a Subset of PEDISTAD Patients
Brief Title: A Study to Assess the Reliability/Feasibility of Using Emerald Touchless Sensor for Scratching and Sleep Quantification in a Subset of Participants From PEDISTAD Study (OBS15333; NCT03687359)
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: LPS17339; U1111-1269-6688 (Registry Identifier: ICTRP)
Record Dates: First submitted 2022-02-01; First posted 2022-02-11 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Dermatitis Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subset of study-OBS15333 patients: As a sub-study of the OBS15333 pediatric AD registry (PEDISTAD), all participants in this study will be receiving standard care of therapies for moderate to severe AD.

SUMMARY:
Primary objective: To explore and quantify the association between nighttime scratching and sleep patterns objectively in pediatric participants with moderate to severe atopic dermatitis (AD) using an innovative Emerald touchless sensor.

Secondary objective: To evaluate the feasibility of using the Emerald touchless sensor in a pediatric clinical trial setting.

DETAILED DESCRIPTION:
16 weeks

ELIGIBILITY:
Inclusion Criteria:

* Participation in OBS15333 pediatric AD registry (PEDISTAD) in the United States (US) study sites.
* Enrolled in PEDISTAD, age more than or equal to 6 years to less than 12 years at the time of enrollment.
* Peak pruritus Numeric Rating Scale (NRS) last night more than or equal to 4 at screening.
* Participant must have home access to reliable and operational Wi-Fi and broadband internet at screening and throughout the study period.
* Participants/parents must have a device (mobile phone, tablet or computer) to record daily itch and sleep disturbance at screening and throughout the study period.
* Participant agrees to sleep by himself/herself (ie, with no other individuals or pets) in the monitored bedroom for the duration of the study (if not all times, at least 5 days a week for a minimum of 5 hours/night for a total of 16 weeks).
* Signed informed consent by the parent/legally acceptable representative and assent by the participant appropriate to the participant's age.

Exclusion Criteria:

- Known history of a childhood sleep disorder such as parasomnias (sleep walking, talking, terrors, etc.), behavioral insomnia of childhood, or restless leg syndrome.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Only participants enrolled in the OBS15333 pediatric AD registry (PEDISTAD) in the United States (US) study sites will be allowed to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
Correlation between weekly averages of Emerald nightly scratching events/hour and Emerald derived sleep efficiency | Week -1 (baseline) to week 12
  Total no. of scratching events and scratching duration within each sleep stage each night will be calculated. Sleep efficiency: total time spent in a sleep stage (Stage 2, 3 or Rapid Eye Movement (REM) stage) relative to the total time in bed will be expressed as a %. Total time in bed: time from when the person enters the bed area and they become relatively static to waking up for the day. Correlation coefficient will be derived using data pairs from baseline through 12 weeks using evaluable data.

SECONDARY OUTCOMES:
Percentage (%) of nights with unusable data | Week -1 (baseline) to week 12
  The weekly average values (both baseline and post baseline, Emerald and participant reported) will be considered evaluable if they are based on at least 3 evaluable nightly values. Nights with unusable Emerald data are defined as nights with no data being collected by the device for any reason or the data collected were unevaluable.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- United States (7):
  - C2 Research Center, LLC-Site Number:8400071, Montgomery, Alabama
  - Amedica Research Institute, Inc.-Site Number:8400067, Hialeah, Florida
  - Eastern Research, Inc.-Site Number:8400032, Hialeah, Florida
  - Skin Research of South Florida, LLC-Site Number:8400018, Miami, Florida
  - Michigan Dermatology Institute-Site Number:8400059, Waterford, Michigan
  - Cincinnati Children's Hospital Medical Center-Site Number:8400017, Cincinnati, Ohio
  - Medical University of South Carolina-Site Number:8400013, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org